CLINICAL TRIAL: NCT04165343
Title: Evaluation of Multi-Organ Metabolism and Perfusion in NAFLD by Total Body Dynamic PET Scan on EXPLORER
Acronym: EXPLORER
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Souvik Sarkar, MD, PhD, Assistant Professor, University of California, Davis
Other Study IDs: 1371653
Record Dates: First submitted 2019-11-06; First posted 2019-11-15 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease (NAFLD); Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Imaging; Echocardiography; Electrocardiography; Caves; Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will order laboratory blood tests as part of this research study and up to 3 tablespoons of blood will be collected for routine clinical and other laboratory tests relevant to the study. An extra of up to 4 teaspoons of blood will be collected for DNA and liver molecules that give information, for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Alcoholic Fatty Liver Disease (NAFLD): Cohort: Patients with known Non-Alcoholic Fatty Liver Disease (NAFLD)
  All patients will undergo the following interventions:
  Positron Emission Tomography (PET) on the EXPLORER scanner Magnetic Resonance Imaging (MRI) Echocardiogram and Electrocardiogram Blood test
  Interventions: Radiation: Positron Emission Tomography (PET) on EXPLORER; Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Echocardiogram and Electrocardiogram; Diagnostic Test: Blood test
- Healthy Control Subjects: Cohort: Healthy controls
  All healthy subjects will undergo the following interventions:
  Positron Emission Tomography (PET) on the EXPLORER scanner Magnetic Resonance Imaging (MRI) Echocardiogram and Electrocardiogram Blood tests
  Interventions: Radiation: Positron Emission Tomography (PET) on EXPLORER; Diagnostic Test: Magnetic Resonance Imaging; Diagnostic Test: Echocardiogram and Electrocardiogram; Diagnostic Test: Blood test

INTERVENTIONS:
Radiation: Positron Emission Tomography (PET) on EXPLORER — Positron Emission Tomography (PET): Your blood sugar level will be checked by a finger stick before the PET scan. A small amount of radioactive "tracer" (approximately 0.5 teaspoons) will be injected into a vein in your arm before the imaging test. You will be asked to lay on your back on the EXPLORER scanner platform with both of your arms over the head during the duration of the test. A small amount of blood (1 tablespoon) will be collected after the test. This test will last for up to one (1) hour. This is a research test. Although the results may be available it cannot be used for clinical care. If any incidental findings are noted, it will be reported to you.
  Other Names: PET Scan
Diagnostic Test: Magnetic Resonance Imaging — MRI will be performed that can measure both the liver stiffness or fibrosis by a method called MR elastography (MRE) and the amount of fat deposited in the liver by MR proton density fat fraction (MR-PDFF). You will be asked to lay on your back on the scanner platform with both of your arms over the head during the duration of the test. MRE and MRI-PDFF are Food and Drugs Administration (FDA) approved tests and the results will be available to you. This test will last up to one (1) hour.
  Other Names: MRI
Diagnostic Test: Echocardiogram and Electrocardiogram — You will have baseline echocardiogram images and electrocardiogram (ECG) taken and will be asked to walk on a treadmill, which will increase in elevation and speed every 3 minutes until you can go no longer. This usually takes 9 to 12 minutes. Immediately after exercise, echocardiogram images and ECG will be taken again. The total time you will be in the stress lab including prep time and recovery is about 60 minutes. Wear comfortable or exercise clothing and walking/running shoes. You will be asked to not eat or drink (except for water) for 4 hours prior to the time of your test. Please drink water the day of the test so you are not dehydrated. This is an FDA approved test and the results will be available to you.
  Other Names: Echo and EKG or ECG
Diagnostic Test: Blood test — We will order laboratory blood tests as part of this research study and up to 3 tablespoons of blood will be collected for routine clinical and other laboratory tests relevant to the study. If you are able to become pregnant, you will have a urine pregnancy test before you begin the study.
  Other Names: Lab test

SUMMARY:
Evaluation of Multi-Organ Metabolism and Perfusion in Non-Alcoholic Fatty Liver Disease (NAFLD) by Total Body Dynamic PET Scan on EXPLORER

DETAILED DESCRIPTION:
You are invited to participate in a research study that seeks to understand the effect of non-alcoholic fatty liver disease (NAFLD) on organs other than the liver. One of the most common organs affected in patients with NAFLD is the heart. We expect to have about 88 people participate in this study at University of California (UC), Davis. About three-fourths (66) of the participants will be patients who have been diagnosed with NAFLD. The other one-fourth (22) will be healthy individuals with no known liver disease. These healthy subjects will allow researchers to compare healthy organs or body functions with those of persons with NAFLD. The healthy participants are called the "Healthy Control" group. All participants will undergo the same testing.

If you agree to participate in this study, researchers will first interview you and review your medical records in order to document your medical (clinical) history. You will also have a physical examination by a doctor and a blood test. You will then undergo a series of imaging tests to determine the status of your liver, heart and other internal organs.

All participants will have a PET/CT Scan (Positron Emission Tomography), and an MRI (Magnetic Resonance Imaging). All participants will also have an Electrocardiogram and an Echocardiogram. All Electrocardiogram tests are the same, but there are two types of Echocardiogram tests. One is like a standard ultra-sound imaging of your heart. The other is a "Stress Cardio" that will require you to increase your heart rate on a treadmill before the ultra-sound test. Your study doctor will determine which test you have.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of 18 years and older
2. NAFLD patients with diagnosis of non-alcoholic fatty liver disease will be eligible for enrollment or healthy controls without any history of fatty liver disease or risks association with fatty liver will be eligible

Exclusion Criteria:

1. History of other liver diseases including viral hepatitis B or C (except those cured > 3 years), autoimmune hepatitis, cholestatic diseases, significant alcohol use or known alcoholic liver disease
2. Participation in a blinded investigational study for NAFLD
3. Pregnant women
4. Prisoners
5. Claustrophobic to MRI and/or PET Scan (EXPLORER)
6. Inability to lie or to maintain posture in the scanner for one hour
7. Hgb A1c >9%
8. Underwent dynamic FDG PET as part of another study, Non-Invasive Evaluation of Liver Steatosis, Inflammation and Fibrosis (IRB 840422) within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Individuals of 18 years and older
  2. NAFLD patients with diagnosis of non-alcoholic fatty liver disease will be eligible for enrollment or healthy controls without any history of fatty liver disease or risks association with fatty liver will be eligible
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Change in myocardial glucose uptake rate (K1) in patient with stage 3-4 liver fibrosis relative to stage 0-2 liver fibrosis | 3 years total study period. Fluorodeoxyglucose (FDG) PET scan study is for 60 minutes.
  The primary outcome is to determine heart (myocardial) glucose uptake rate (K1) determined by dynamic FDG PET scan. This will be compared between those with liver fibrosis stage 3-4 with those with lower stage of fibrosis stage 0-2 as determined by magnetic resonance elastography.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No